CLINICAL TRIAL: NCT02219256
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Safety, Tolerability and Pharmacokinetic Study of Escalating Single Intravenous Infusion and Subcutaneous Administration of TAK-079 in Healthy Subjects
Brief Title: A Phase 1 Study to Assess the Safety, Tolerability, and Pharmacokinetics of TAK-079 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-079_101; U1111-1155-5857 (Registry Identifier: WHO); 2013-004210-18 (EudraCT Number); 14/LO/1070 (Registry Identifier: NRES)
Record Dates: First submitted 2014-08-14; First posted 2014-08-18 (Estimated); Results first posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-03

CONDITIONS: Autoimmune Disease
Keywords: Drug therapy
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1: TAK-079 0.0003 mg/kg (Experimental): TAK-079 0.0003 mg/kg, infusion, intravenously, once.
  Interventions: Drug: TAK-079
- Cohort 2-9: TAK-079 TBD (Experimental): TAK-079, infusion, intravenously or subcutaneously, once. Dose to be determined from data collected in previous IV or SC Cohort(s)
  Interventions: Drug: TAK-079
- Placebo to TAK-079 (Placebo Comparator): Placebo to TAK-079, infusion, intravenously or subcutaneously, once.
  Interventions: Drug: Placebo to TAK-079

INTERVENTIONS:
Drug: TAK-079 — TAK-079 solution
  Arms: Cohort 1: TAK-079 0.0003 mg/kg; Cohort 2-9: TAK-079 TBD
Drug: Placebo to TAK-079 — Placebo to TAK-079 solution
  Arms: Placebo to TAK-079

SUMMARY:
The purpose of this study is to characterize the pharmacokinetic and safety and tolerability profile of TAK-079 following a single intravenous (IV) infusion or subcutaneous (SC) administration at escalating dose levels in healthy participants.

DETAILED DESCRIPTION:
The drug being tested in this study is TAK-079. TAK-079 is being tested to find a safe and well-tolerated dose and to assess how TAK-079 is processed by the body. This study will look at pharmacokinetics, side effects, and laboratory results in people who take TAK-079 and is designed as a randomized single dose-rising study.

Therefore, each subsequent cohort will not start until the previous cohort has completed and the results are reviewed. Each participant will receive TAK-079 or placebo once only as an IV infusion or by SC administration. The starting dose for IV will be 0.0003 mg/kg and SC dose of 0.01 or 0.03 mg/kg was determined based on the no-observed-adverse-effect-level (NOAEL) results from the 13-week good laboratory practice (GLP) monkey toxicology study. If this dose is well-tolerated, the next group will receive a higher dose, etc, until a maximal tolerated dose is reached with the highest dose not to exceed 1.0 mg/kg.

This single-center trial will be conducted in the United Kingdom. The overall time to participate in this study is up to 17 weeks. Participants will make 11 visits to the clinic, including one 10-day period of confinement in the clinic. All participants will be contacted by telephone 14 days after the last visit to the clinic for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy male or female with no child bearing potential who is 18 to 55 years of age inclusive.
2. The subject weighs at least 70 kilogram (kg) for cohort 1 and subsequent cohorts 50 kg (110.2 lb) and less than 100 kg (220.5 lb) and has a body mass index (BMI) range of 18.5 to 30 kilogram per square meter (kg/m^2), inclusive at Screening Visit 1.
3. A male participant who is non-sterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 6 months after last dose of study medication.

Exclusion Criteria:

1. Has received any investigational compound within the last 3 months or 5*T1/2 of the investigational compound,whichever is longer, prior to the day of study medication (Day 1).
2. Has received any live vaccinations, within the last 3 months prior to Screening or is expected to receive any vaccinations during the study or for 1 month after the Day 78 Study Exit visit.
3. Has received any other biologic medical products at any time in the past.
4. Has a positive drug or alcohol screening result, or a history of drug or alcohol abuse.
5. Has a positive test result for hepatitis or human immunodeficiency virus antibody.
6. Has any signs of an acute infection or history of frequent or chronic infection, or herpes zoster.
7. Has active or latent tuberculosis (TB)
8. Considered unfit for the study by the Principal Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2014-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (2):
- United Kingdom (2):
  - London, London
  - Headington, Oxford

REFERENCES:
- [Derived] Fedyk ER, Zhao L, Koch A, Smithson G, Estevam J, Chen G, Lahu G, Roepcke S, Lin J, Mclean L. Safety, tolerability, pharmacokinetics and pharmacodynamics of the anti-CD38 cytolytic antibody TAK-079 in healthy subjects. Br J Clin Pharmacol. 2020 Jul;86(7):1314-1325. doi: 10.1111/bcp.14241. Epub 2020 Feb 22. PMID 32045493

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United Kingdom (UK) from 01 August 2014 to 29 April 2016.
Pre-assignment Details: Healthy participants were enrolled in 1 of 12 treatment groups to receive: TAK-079 placebo, 0.0003, 0.001, 0.003, 0.01, 0.03, 0.06 milligram per kilogram (mg/kg) Intravenously (IV) and TAK-079 placebo, 0.03, 0.1, 0.3, 0.6 mg/kg subcutaneously (SC).
Groups:
- TAK-079 Pooled Placebo IV: TAK-079 placebo-matching, infusion solution, IV, once on Day 1.
- TAK-079 0.0003 mg/kg IV: TAK-079 0.0003 mg/kg, infusion solution, IV, once on Day 1.
- TAK-079 0.001 mg/kg IV: TAK-079 0.001 mg/kg, infusion solution, IV, once on Day 1.
- TAK-079 0.003 mg/kg IV: TAK-079 0.003 mg/kg, infusion solution, IV, once on Day 1.
- TAK-079 0.01 mg/kg IV: TAK-079 0.01 mg/kg, infusion solution, IV, once on Day 1.
- TAK-079 0.03 mg/kg IV: TAK-079 0.03 mg/kg, infusion solution, IV, once on Day 1.
- TAK-079 0.06 mg/kg IV: TAK-079 0.06 mg/kg, infusion solution, IV, once on Day 1.
- TAK-079 Pooled Placebo SC: TAK-079 placebo-matching, infusion solution, SC, once on Day 1.
- TAK-079 0.03 mg/kg SC: TAK-079 0.03 mg/kg, infusion solution, SC, once on Day 1.
- TAK-079 0.1 mg/kg SC: TAK-079 0.01 mg/kg, infusion solution, SC, once on Day 1
- TAK-079 0.3 mg/kg SC: TAK-079 0.3 mg/kg, infusion solution, SC, once on Day 1.
- TAK-079 0.6 mg/kg SC: TAK-079 0.6 mg/kg, infusion solution, SC, once on Day 1.
Period: Overall Study
Arm/Group | TAK-079 Pooled Placebo IV | TAK-079 0.0003 mg/kg IV | TAK-079 0.001 mg/kg IV | TAK-079 0.003 mg/kg IV | TAK-079 0.01 mg/kg IV | TAK-079 0.03 mg/kg IV | TAK-079 0.06 mg/kg IV | TAK-079 Pooled Placebo SC | TAK-079 0.03 mg/kg SC | TAK-079 0.1 mg/kg SC | TAK-079 0.3 mg/kg SC | TAK-079 0.6 mg/kg SC
Started | 12 | 4 | 4 | 4 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6
Completed | 12 | 4 | 4 | 4 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were enrolled, received 1 dose of study drug (after study drug dosing started) including those who did not complete all scheduled study visits.
Groups:
- Total: Total of all reporting groups
Arm/Group | TAK-079 Pooled Placebo IV | TAK-079 0.0003 mg/kg IV | TAK-079 0.001 mg/kg IV | TAK-079 0.003 mg/kg IV | TAK-079 0.01 mg/kg IV | TAK-079 0.03 mg/kg IV | TAK-079 0.06 mg/kg IV | TAK-079 Pooled Placebo SC | TAK-079 0.03 mg/kg SC | TAK-079 0.1 mg/kg SC | TAK-079 0.3 mg/kg SC | TAK-079 0.6 mg/kg SC | Total
Number analyzed (Participants) | 12 | 4 | 4 | 4 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (10.61) | 23.5 (3.42) | 42.3 (12.12) | 32.8 (10.72) | 36.2 (9.52) | 32.3 (5.92) | 35.7 (11.60) | 34.9 (13.61) | 36.7 (10.33) | 31.0 (8.15) | 40.8 (7.83) | 27.7 (8.16) | 34.3 (10.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Male | 12 | 4 | 4 | 4 | 6 | 6 | 6 | 7 | 6 | 6 | 6 | 6 | 73
Race/Ethnicity, Customized [Number; unit: participants]
  White | 8 | 3 | 2 | 3 | 4 | 5 | 5 | 6 | 4 | 3 | 6 | 2 | 51
  Black or African American | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 4
  Asian | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 3 | 0 | 3 | 13
  Multiracial | 1 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 6
Region of Enrollment [Number; unit: participants]
  United Kingdom | 12 | 4 | 4 | 4 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 74
Smoking Classification [Number; unit: participants]
  Currently smoking | 4 | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 1 | 1 | 1 | 1 | 13
  Never smoked | 6 | 2 | 2 | 3 | 3 | 2 | 4 | 7 | 3 | 4 | 4 | 4 | 44
  Ex-smoker | 2 | 2 | 1 | 1 | 2 | 1 | 2 | 1 | 2 | 1 | 1 | 1 | 17
Caffeine Classification [Number; unit: participants]
  Had caffeine consumption | 9 | 3 | 3 | 1 | 6 | 6 | 3 | 3 | 3 | 6 | 5 | 2 | 50
  Had no caffeine consumption | 3 | 1 | 1 | 3 | 0 | 0 | 3 | 5 | 3 | 0 | 1 | 4 | 24
Alcohol Classification [Number; unit: participants]
  Drinks everyday | 5 | 1 | 2 | 1 | 3 | 1 | 4 | 2 | 4 | 1 | 2 | 4 | 30
  Never drank | 7 | 3 | 2 | 3 | 3 | 5 | 2 | 6 | 2 | 5 | 4 | 2 | 44
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 174.7 (9.17) | 181.3 (6.90) | 175.0 (8.04) | 179.5 (10.91) | 173.8 (1.47) | 175.5 (7.97) | 173.8 (7.03) | 177.8 (7.91) | 176.8 (3.31) | 181.2 (8.80) | 177.8 (6.68) | 172.3 (4.32) | 176.3 (7.32)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 73.98 (7.355) | 80.63 (8.768) | 76.68 (9.011) | 72.10 (9.090) | 75.45 (11.042) | 69.12 (8.043) | 71.32 (6.187) | 78.53 (12.508) | 79.77 (8.584) | 75.18 (9.887) | 79.73 (8.311) | 71.25 (9.434) | 75.20 (9.149)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 24.32 (2.507) | 24.53 (2.337) | 25.05 (2.456) | 22.33 (1.176) | 24.93 (3.420) | 22.45 (2.118) | 23.60 (1.383) | 24.80 (3.311) | 25.52 (2.763) | 22.85 (1.947) | 25.22 (2.225) | 23.98 (3.064) | 24.18 (2.553)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience at Least 1 Treatment-emergent Adverse Event (TEAE) and Serious Adverse Event (SAE)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug. AE was assessed according to severity; mild (transient and easily tolerated by the participant), moderate (causes the participant discomfort and interrupts the participant's usual activities) and severe (causes considerable interference with the participant's usual activities).
Time Frame: First dose up to Day 94
Population: The safety analysis set included all participants who were enrolled, received 1 dose of study drug (after study drug dosing started) inclusive of those participants who did not complete all scheduled study visits.
Measure: Number; unit: participants
Arm/Group | TAK-079 Pooled Placebo IV | TAK-079 0.0003 mg/kg IV | TAK-079 0.001 mg/kg IV | TAK-079 0.003 mg/kg IV | TAK-079 0.01 mg/kg IV | TAK-079 0.03 mg/kg IV | TAK-079 0.06 mg/kg IV | TAK-079 Pooled Placebo SC | TAK-079 0.03 mg/kg SC | TAK-079 0.1 mg/kg SC | TAK-079 0.3 mg/kg SC | TAK-079 0.6 mg/kg SC
Number analyzed (Participants) | 12 | 4 | 4 | 4 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6
participants
  TEAE: Mild | 6 | 3 | 2 | 1 | 5 | 4 | 2 | 3 | 5 | 4 | 4 | 4
  TEAE: Moderate | 5 | 0 | 1 | 2 | 1 | 2 | 4 | 3 | 1 | 2 | 1 | 1
  TEAE: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Who Meet the Takeda Development Centre (TDC) Markedly Abnormal Criteria for Safety Laboratory Tests at Least Once Post Dose
Time Frame: First dose up to Day 78
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | TAK-079 Pooled Placebo IV | TAK-079 0.0003 mg/kg IV | TAK-079 0.001 mg/kg IV | TAK-079 0.003 mg/kg IV | TAK-079 0.01 mg/kg IV | TAK-079 0.03 mg/kg IV | TAK-079 0.06 mg/kg IV | TAK-079 Pooled Placebo SC | TAK-079 0.03 mg/kg SC | TAK-079 0.1 mg/kg SC | TAK-079 0.3 mg/kg SC | TAK-079 0.6 mg/kg SC
Number analyzed (Participants) | 12 | 4 | 4 | 4 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6
participants | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2

3. Secondary Outcome: Cmax: Maximum Observed Serum Concentration for TAK-079
Time Frame: Day 1 pre-dose and at multiple time-points (up to Day 78) post-dose
Population: The pharmacokinetic(PK) analysis set included all participants who received study drug and had at least 1 measurable serum concentration of TAK-079. PK analysis was performed for TAK-079 0.03, 0.06 mg/kg IV and 0.6 SC mg/kg dose groups only, since serum concentrations of TAK-079 were below the LLOQ at all PK sampling time-points for remaining arms.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | TAK-079 Pooled Placebo IV | TAK-079 0.0003 mg/kg IV | TAK-079 0.001 mg/kg IV | TAK-079 0.003 mg/kg IV | TAK-079 0.01 mg/kg IV | TAK-079 0.03 mg/kg IV | TAK-079 0.06 mg/kg IV | TAK-079 Pooled Placebo SC | TAK-079 0.03 mg/kg SC | TAK-079 0.1 mg/kg SC | TAK-079 0.3 mg/kg SC | TAK-079 0.6 mg/kg SC
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 0 | 0 | 0 | 0 | 5
nanogram per milliliter (ng/mL) |  |  |  |  |  | 21.4 (8.3) | 100.4 (51.7) |  |  |  |  | 23.0 (15.5)

4. Secondary Outcome: AUClast: Area Under the Serum Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-079
Time Frame: Day 1 pre-dose and at multiple time points (up to Day 78) post-dose
Population: The PK analysis set:all participants who received study drug and had at least 1 measurable serum concentration of TAK-079.A valid AUClast was derived for TAK-079 0.6 mg/kgSC dose group only, since serum concentrations of TAK-079 were either below the LLOQ at all PK sampling time-points or too limited to estimate AUClast reliably for remaining arms.
Measure: Mean (Standard Deviation); unit: nanogram*day per milliliter (ng*day/mL)
Arm/Group | TAK-079 Pooled Placebo IV | TAK-079 0.0003 mg/kg IV | TAK-079 0.001 mg/kg IV | TAK-079 0.003 mg/kg IV | TAK-079 0.01 mg/kg IV | TAK-079 0.03 mg/kg IV | TAK-079 0.06 mg/kg IV | TAK-079 Pooled Placebo SC | TAK-079 0.03 mg/kg SC | TAK-079 0.1 mg/kg SC | TAK-079 0.3 mg/kg SC | TAK-079 0.6 mg/kg SC
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
nanogram*day per milliliter (ng*day/mL) |  |  |  |  |  |  |  |  |  |  |  | 90.4 (83.2)

5. Secondary Outcome: AUC∞: Area Under the Serum Concentration-time Curve From Time 0 to Infinity for TAK-079
Time Frame: Day 1 pre-dose and at multiple time-points (up to Day 78) post-dose
Population: The PK analysis set included all participants who received study drug and had at least 1 measurable serum concentration of TAK-079. PK analysis was performed for TAK-079 0.6 mg/kg SC dose groups only, since serum concentrations of TAK-079 were below the LLOQ at all PK sampling time-points for remaining arms.
Measure: Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | TAK-079 Pooled Placebo IV | TAK-079 0.0003 mg/kg IV | TAK-079 0.001 mg/kg IV | TAK-079 0.003 mg/kg IV | TAK-079 0.01 mg/kg IV | TAK-079 0.03 mg/kg IV | TAK-079 0.06 mg/kg IV | TAK-079 Pooled Placebo SC | TAK-079 0.03 mg/kg SC | TAK-079 0.1 mg/kg SC | TAK-079 0.3 mg/kg SC | TAK-079 0.6 mg/kg SC
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
ng*day/mL |  |  |  |  |  |  |  |  |  |  |  | 212 (103)

6. Secondary Outcome: Percentage of Participants With Positive Antidrug Antibody (ADA) and Neutralizing Antibody (Nab)
Description: Results for ADA analysis were reported.
Time Frame: Baseline up to Day 78
Population: The safety analysis set included all participants who were enrolled, received 1 dose of study drug (after study drug dosing started) inclusive of those participants who did not complete all scheduled study visits. Due to change in planned analysis testing of NAb activity of ADA positive samples was not analysed.
Measure: Number; unit: percentage of participants
Arm/Group | TAK-079 Pooled Placebo IV | TAK-079 0.0003 mg/kg IV | TAK-079 0.001 mg/kg IV | TAK-079 0.003 mg/kg IV | TAK-079 0.01 mg/kg IV | TAK-079 0.03 mg/kg IV | TAK-079 0.06 mg/kg IV | TAK-079 Pooled Placebo SC | TAK-079 0.03 mg/kg SC | TAK-079 0.1 mg/kg SC | TAK-079 0.3 mg/kg SC | TAK-079 0.6 mg/kg SC
Number analyzed (Participants) | 12 | 4 | 4 | 4 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 33.3 | 16.7 | 0 | 16.7 (102.58826)

7. Primary Outcome: Number of Participants Who Meet the TDC Markedly Abnormal Criteria for Vital Sign Measurements at Least Once Post Dose
Time Frame: First dose up to Day 78
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | TAK-079 Pooled Placebo IV | TAK-079 0.0003 mg/kg IV | TAK-079 0.001 mg/kg IV | TAK-079 0.003 mg/kg IV | TAK-079 0.01 mg/kg IV | TAK-079 0.03 mg/kg IV | TAK-079 0.06 mg/kg IV | TAK-079 Pooled Placebo SC | TAK-079 0.03 mg/kg SC | TAK-079 0.1 mg/kg SC | TAK-079 0.3 mg/kg SC | TAK-079 0.6 mg/kg SC
Number analyzed (Participants) | 12 | 4 | 4 | 4 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6
participants | 6 | 2 | 2 | 2 | 1 | 4 | 6 | 4 | 4 | 4 | 3 | 1

8. Primary Outcome: Number of Participants Who Meet the TDC Markedly Abnormal Criteria for Safety 12-lead Electrocardiogram (ECG) Parameters at Least Once Post Dose
Time Frame: First dose up to Day 78
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | TAK-079 Pooled Placebo IV | TAK-079 0.0003 mg/kg IV | TAK-079 0.001 mg/kg IV | TAK-079 0.003 mg/kg IV | TAK-079 0.01 mg/kg IV | TAK-079 0.03 mg/kg IV | TAK-079 0.06 mg/kg IV | TAK-079 Pooled Placebo SC | TAK-079 0.03 mg/kg SC | TAK-079 0.1 mg/kg SC | TAK-079 0.3 mg/kg SC | TAK-079 0.6 mg/kg SC
Number analyzed (Participants) | 12 | 4 | 4 | 4 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6
participants | 8 | 3 | 3 | 1 | 3 | 5 | 1 | 5 | 4 | 5 | 1 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 94 days after the last dose of double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-079 Pooled Placebo IV | TAK-079 0.0003 mg/kg IV | TAK-079 0.001 mg/kg IV | TAK-079 0.003 mg/kg IV | TAK-079 0.01 mg/kg IV | TAK-079 0.03 mg/kg IV | TAK-079 0.06 mg/kg IV | TAK-079 Pooled Placebo SC | TAK-079 0.03 mg/kg SC | TAK-079 0.1 mg/kg SC | TAK-079 0.3 mg/kg SC | TAK-079 0.6 mg/kg SC
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/4 | 0/4 | 0/4 | 0/6 | 0/6 | 0/6 | 0/8 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 11/12 | 3/4 | 3/4 | 3/4 | 6/6 | 6/6 | 6/6 | 6/8 | 6/6 | 6/6 | 5/6 | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-079 Pooled Placebo IV (N=12) | TAK-079 0.0003 mg/kg IV (N=4) | TAK-079 0.001 mg/kg IV (N=4) | TAK-079 0.003 mg/kg IV (N=4) | TAK-079 0.01 mg/kg IV (N=6) | TAK-079 0.03 mg/kg IV (N=6) | TAK-079 0.06 mg/kg IV (N=6) | TAK-079 Pooled Placebo SC (N=8) | TAK-079 0.03 mg/kg SC (N=6) | TAK-079 0.1 mg/kg SC (N=6) | TAK-079 0.3 mg/kg SC (N=6) | TAK-079 0.6 mg/kg SC (N=6)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site bruise (General disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site phlebitis (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site related reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Instillation site bruise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 3 | 1 | 3
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epididymitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 0 | 0 | 1 | 2 | 3 | 5 | 2 | 2 | 1 | 1 | 3
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 1 | 0 | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Initial insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 0 | 1 | 1
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.